CLINICAL TRIAL: NCT00911651
Title: Open, Randomized, Two-Way Crossover, Pilot Study to Assess the Effect of Salbutamol in Comparison With Ipratropium Bromide on Central and Peripheral Airway Dimensions in COPD Patients
Brief Title: Study to Assess the Effect of Salbutamol and Ipratropium Bromide in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Prof Wilfried De Backer, Antwerp University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PML_DOC_0801
Record Dates: First submitted 2009-05-28; First posted 2009-06-02 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-05

CONDITIONS: COPD
Keywords: COPD; salbutamol; ipratropium bromide; computational fluid dynamics; functional imaging; central and peripheral airways
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Ipratropium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- salbutamol (Active Comparator): 6 patients with moderate (GOLD 2) and severe (GOLD 3) COPD
  Interventions: Drug: Salbutamol
- ipratropium bromide (Active Comparator): COPD patients GOLD stage II and III
  Interventions: Drug: ipratropium bromide

INTERVENTIONS:
Drug: Salbutamol — 400 µg inhalation once
  Other Names: Ventolin
  Arms: salbutamol
Drug: ipratropium bromide — 80 µg inhalation once
  Other Names: atrovent
  Arms: ipratropium bromide

SUMMARY:
The objectives of this study are to assess the effect of salbutamol in comparison with ipratropium bromide on the geometry of central and peripheral airways and to correlate spirometric indices with the Computational Fluid Dynamics (CFD) based calculated airway volumes and resistances for both compounds.

DETAILED DESCRIPTION:
Salbutamol (VentolinTM) is a short acting beta agonist (SABA) which is used to treat wheezing, dyspnea and breathing difficulties caused by asthma and COPD. Further, it is also used to prevent bronchospasm during exercise.

Ipratropium bromide (Atrovent® HFA) is a short acting anticholinergic bronchodilator (short acting muscarinic antagonist (SAMA)) that improves lung function, dyspnea, exercise tolerance and health-related quality of life in patients with COPD. Studies have also shown that ipratropium bromide might reduce COPD exacerbations and related hospitalisations because the extended bronchodilatation might reduce infection rates by improving clearance of respiratory secretions.

In this open, randomized, two-way crossover, pilot study the effect of salbutamol in patients with moderate and severe COPD will be examined in comparison with the effects of ipratropium bromide. These patients will receive 400 µg salbutamol and 80 µg ipratropium bromide in a randomized crossover design.

The objectives of this study are to assess the effect of salbutamol in comparison with ipratropium bromide on the geometry of central and peripheral airways and to correlate spirometric indices (as Forced Expiratory Volume in one second (FEV1) and Tiffeneau index) with the Computational Fluid Dynamics (CFD) based calculated airway volumes and resistances for both compounds.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented COPD based on the following criteria:

   * Smoking history of at least 10 pack-years.
   * Decreased Tiffeneau index (FEV1/(F)VC < 0.70).
2. Patients aged ≥ 40 years.
3. Patients should present moderate to severe COPD with an FEV1 between 30 and 80% of predicted (GOLD 2 and 3).
4. Patients should be treated according to GOLD guidelines.
5. Able to inhale study drug.
6. Maintained on stable respiratory medications for 6 weeks prior to visit 1.
7. Able to perform lung function tests.
8. Able to follow study procedures.

Exclusion Criteria:

1. Patients who are allergic to salbutamol, ipratropium bromide or to another element of the product.
2. Patients allergic to sojalecithin and products on the basis of soja and peanut.
3. Patients who have or ever had glaucoma.
4. Patients with urinary problems, prostate hyperplasy or bladder-neck obstruction. Patients whose symptoms are controlled on treatment may be included.
5. Patients with a recent history (i.e. six months or less) of myocardial infarction.
6. Patients with any unstable or life threatening cardiac arrhythmia.
7. Patients with severe kidney insufficiency (creatinine clearance ≤50 ml/min)a.
8. Patients below the age of 40.
9. Patients who are pregnant or are breast-feeding.
10. Patients who are treated with other anticholinergic medications, that cannot be stopped during the study period.
11. A respiratory infection or exacerbation of COPD in the four weeks prior to screening.
12. Significant alcohol or drug abuse within the past 12 months.
13. Participation in another trial with an investigational drug within one month or six half lives (whichever is greater) prior to screening visit.
14. Known active tuberculosis.
15. A history of asthma, cystic fibrosis, central bronchiectasis, interstitial lung disease or pulmonary thromboembolic disease.
16. A history of thoracotomy with pulmonary resection.
17. Active or untreated malignancy.
18. Use of oral corticosteroid medication at unstable doses (i.e. less than six weeks on a stable dose) or at doses ≥ 10 mg/day.

a Cockroft's formulae should be applied: in male: creatinine clearance = (140-age) x weight / 72 x creatininemia in female: creatinine clearance = 0.85 x (140-age) x weight / 72 x creatininemia

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the effect of a single dose of salbutamol in comparison with ipratropium bromide on central and peripheral small airways with high-resolution/multislice CT scan imaging technique. | 1 month

SECONDARY OUTCOMES:
The secondary objectives are to evaluate effects on spirometric indices to correlate these with the CFD based calculated airway volumes and resistances for both compounds and to evaluate the safety of the products. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried A De Backer, MD PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Antwerp, Antwerp, Belgium